CLINICAL TRIAL: NCT07270302
Title: Safety and Efficacy of Nebulized Nasal Steroids for the Treatment of Chronic Rhinosinusitis
Brief Title: Nebulized Nasal Steroids
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202503084
Record Dates: First submitted 2025-11-25; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Chronic Rhinosinusitis
Keywords: Otolaryngology; Pharmacology; Pharmacy; intranasal steroid sprays

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Study coordinators will be blinded to treatment arm during data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- nebulizer group (Experimental): Subjects in the nebulizer group will be prescribed a 42-day supply of 0.5 mg budesonide packets, to be used twice daily without any concomitant saline lavage.
  Interventions: Combination Product: nebulized budesonide via NasoNeb
- budesonide lavage group (Active Comparator): Subjects in the budesonide lavage group will be prescribed 42-day supply of 0.5 mg budesonide packets to be administered via 240 mL twice daily nasal saline lavage.
  Interventions: Combination Product: budesonide lavage via NeilMed

INTERVENTIONS:
Combination Product: nebulized budesonide via NasoNeb — For the nebulization group, each dose will be dissolved in 10 mL saline with 5 mL nebulized solution being applied to each nasal cavity.
  Device: NasoNeb
  Arms: nebulizer group
Combination Product: budesonide lavage via NeilMed — For the lavage group, each dose will be dissolved in 240 mL saline and 120 mL of the solution will be administered to each nasal cavity.
  Device: NeilMed
  Arms: budesonide lavage group

SUMMARY:
The goal of the proposed project is to assess the efficacy, safety, and patient experience of budesonide administered via the NasoNeb system for medical management of CRS. The authors propose a randomized controlled trial of nebulized budesonide via the NasoNeb compared against budesonide lavage.

DETAILED DESCRIPTION:
Chronic rhinosinusitis is primarily an inflammatory disorder affecting up to 1 in 8 individuals and causing economic burden of greater than 13 billion USD. The NasoNeb is FDA approved for the nasal administration of medications; however, it has been scarcely studied in the existing literature. Many patients are intolerant of or non-compliant with other modalities of nasal steroid administration, and the NasoNeb represents a potential new treatment method for these patients.

Participants will be provided with either a NasoNeb machine or NeilMed lavage bottle, and a prescription for a 42-day supply of 0.5 mg budesonide packets, to be used twice daily. For the NasoNeb, each dose will be dissolved in 10 mL saline with 5 mL nebulized solution being applied to each nasal cavity. This dose was chosen given the historical evidence of efficacy of budesonide 0.5mg daily application via saline lavage.

For the lavage, each budesonide dose will be dissolved in 240 mL saline. Participants will be shown proper use of the NasoNeb machine or lavage bottle at the time of enrollment and be given written instructions with links to video tutorials.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older that meet diagnostic criteria for CRS with or without polyposis as documented by their recruiting physician.
* Diagnostic criteria for CRS will be defined according to EPOS criteria of >12 weeks of 2 of the following subjective symptoms: nasal blockage or obstruction, rhinorrhea, hyposmia, or facial pain/pressure AND objective evidence of CRS on either nasal endoscopy or CT scan

Exclusion Criteria:

* Patients who have previously undergone sinus surgery
* Severe polyposis; defined as Lund Kennedy endoscopy score greater than 1
* Patients who are currently using or who have previously used biologic medications for their nasal polyps. These medications include: dupilumab, omalizumab, mepolizumab, tezepelumab, or depemokimab
* Inability to complete surveys in English
* known comorbid mucociliary disease
* known adrenal disease or other HPA dysfunction
* patients taking oral corticosteroids for other medical conditions
* oral antibiotic administration within 2 weeks of study participation
* a baseline SNOT-22 score less than 9, due to inability to achieve the MCID

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Sino-Nasal Outcome Test (SNOT-22) | week 6
  SNOT-22 is a 22-question survey designed to measure the physical, functional, and emotional consequences of rhinosinusitis. It contains questions regarding symptoms commonly associated with sinonasal disease.
  Subjects rate each question by using a 0-5 point scale with 0=no problem, 1=very mild problem, 2=mild or slight problem, 3=moderate problem, 4=severe problem, 5=problem as bad as it can be. The SNOT-22 total score ranges from a minimum score of 0 to a maximum score of 110, with higher scores representing worse outcome.
  9 point difference in SNOT-22 reduction is defined as the minimally clinically important improvement.

SECONDARY OUTCOMES:
Lund-Kennedy scores | week 6
  Lund-Kennedy scores from nasal endoscopy will be recoded. The original LK system evaluates five components, each graded 0 to 2 for each side of nasal cavity. The score from both sides are summed up and for a total score ranging from 0-20 (10 points per side). Higher scores indicate more severe disease.
  Modified scores will be used.
cosyntropin stimulation | week 6
  Patients from both arms may volunteer for cosyntropin stimulation testing. This will be done to monitor for potential adrenal suppression related to treatment.
  Cosyntropin testing yields a numerical value with units of mcg/dL. We will use a threshold of normal to be greater than or equal to 18 mcg/dL at the 60 minute test.
Clinical Global Impression - Improvement (CGI-I) | week 3 and week 6
  The primary outcome measure will be the rate of responders (as a percentage) to the intervention defined as the number of participants reporting 2 (Moderately Improved), or 3 (Much Improved) in the Clinical Global Impression of Improvement (CGI-I) assessed after 6 weeks of treatment divided by the total number of participants in each study group.
  CGI-I asks subjects to rate their overall response to treatment using a 7-point Likert scale ranging from -3 to 3 ("Much Worse" to "Much Improved"). Participants responding 2 (Moderately Improved), or 3 (Much Improved) to the the CGI-I question "Compared to the start of the study, how would you rate your nasal breathing now", will be defined as responders to treatment.
Sino-Nasal Outcome Test (SNOT-22) | week 3
  SNOT-22 is a 22-question survey designed to measure the physical, functional, and emotional consequences of rhinosinusitis. It contains questions regarding symptoms commonly associated with sinonasal disease.
  Subjects rate each question by using a 0-5 point scale with 0=no problem, 1=very mild problem, 2=mild or slight problem, 3=moderate problem, 4=severe problem, 5=problem as bad as it can be. The SNOT-22 total score ranges from a minimum score of 0 to a maximum score of 110, with higher scores representing worse outcome.
  9 point difference in SNOT-22 reduction is defined as the minimally clinically important improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Nyssa Farrell, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Nyssa Fox Farrell, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tait S, Kallogjeri D, Suko J, Kukuljan S, Schneider J, Piccirillo JF. Effect of Budesonide Added to Large-Volume, Low-pressure Saline Sinus Irrigation for Chronic Rhinosinusitis: A Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2018 Jul 1;144(7):605-612. doi: 10.1001/jamaoto.2018.0667. PMID 29879268
- [Background] Orlandi RR, Kingdom TT, Smith TL, Bleier B, DeConde A, Luong AU, Poetker DM, Soler Z, Welch KC, Wise SK, Adappa N, Alt JA, Anselmo-Lima WT, Bachert C, Baroody FM, Batra PS, Bernal-Sprekelsen M, Beswick D, Bhattacharyya N, Chandra RK, Chang EH, Chiu A, Chowdhury N, Citardi MJ, Cohen NA, Conley DB, DelGaudio J, Desrosiers M, Douglas R, Eloy JA, Fokkens WJ, Gray ST, Gudis DA, Hamilos DL, Han JK, Harvey R, Hellings P, Holbrook EH, Hopkins C, Hwang P, Javer AR, Jiang RS, Kennedy D, Kern R, Laidlaw T, Lal D, Lane A, Lee HM, Lee JT, Levy JM, Lin SY, Lund V, McMains KC, Metson R, Mullol J, Naclerio R, Oakley G, Otori N, Palmer JN, Parikh SR, Passali D, Patel Z, Peters A, Philpott C, Psaltis AJ, Ramakrishnan VR, Ramanathan M Jr, Roh HJ, Rudmik L, Sacks R, Schlosser RJ, Sedaghat AR, Senior BA, Sindwani R, Smith K, Snidvongs K, Stewart M, Suh JD, Tan BK, Turner JH, van Drunen CM, Voegels R, Wang Y, Woodworth BA, Wormald PJ, Wright ED, Yan C, Zhang L, Zhou B. International consensus statement on allergy and rhinology: rhinosinusitis 2021. Int Forum Allergy Rhinol. 2021 Mar;11(3):213-739. doi: 10.1002/alr.22741. PMID 33236525
- [Background] Rudmik L. Economics of Chronic Rhinosinusitis. Curr Allergy Asthma Rep. 2017 Apr;17(4):20. doi: 10.1007/s11882-017-0690-5. PMID 28337570
- [Background] Chung SD, Hung SH, Lin HC, Lin CC. Health care service utilization among patients with chronic rhinosinusitis: a population-based study. Laryngoscope. 2014 Jun;124(6):1285-9. doi: 10.1002/lary.24500. Epub 2013 Dec 10. PMID 24338913
- [Background] Bhattacharyya N. Contemporary assessment of the disease burden of sinusitis. Allergy Rhinol (Providence). 2010 Jan 1;1(1):8. doi: 10.2500/ajra.2009.23.3355. No abstract available. PMID 28569228
- [Background] Bhattacharyya N, Orlandi RR, Grebner J, Martinson M. Cost burden of chronic rhinosinusitis: a claims-based study. Otolaryngol Head Neck Surg. 2011 Mar;144(3):440-5. doi: 10.1177/0194599810391852. Epub 2011 Feb 3. PMID 21493210
- [Background] Phillips KM, Hoehle LP, Bergmark RW, Caradonna DS, Gray ST, Sedaghat AR. Acute Exacerbations Mediate Quality of Life Impairment in Chronic Rhinosinusitis. J Allergy Clin Immunol Pract. 2017 Mar-Apr;5(2):422-426. doi: 10.1016/j.jaip.2016.09.015. Epub 2016 Nov 7. PMID 27839750
- [Background] Phillips KM, Hoehle LP, Caradonna DS, Gray ST, Sedaghat AR. Minimal clinically important difference for the 22-item Sinonasal Outcome Test in medically managed patients with chronic rhinosinusitis. Clin Otolaryngol. 2018 Oct;43(5):1328-1334. doi: 10.1111/coa.13177. Epub 2018 Jul 26. PMID 29953729
- [Background] Stevens WW, Peters AT, Tan BK, Klingler AI, Poposki JA, Hulse KE, Grammer LC, Welch KC, Smith SS, Conley DB, Kern RC, Schleimer RP, Kato A. Associations Between Inflammatory Endotypes and Clinical Presentations in Chronic Rhinosinusitis. J Allergy Clin Immunol Pract. 2019 Nov-Dec;7(8):2812-2820.e3. doi: 10.1016/j.jaip.2019.05.009. Epub 2019 May 22. PMID 31128376
- [Background] Chong LY, Head K, Hopkins C, Philpott C, Burton MJ, Schilder AG. Different types of intranasal steroids for chronic rhinosinusitis. Cochrane Database Syst Rev. 2016 Apr 26;4(4):CD011993. doi: 10.1002/14651858.CD011993.pub2. PMID 27115215
- [Background] Joe SA, Thambi R, Huang J. A systematic review of the use of intranasal steroids in the treatment of chronic rhinosinusitis. Otolaryngol Head Neck Surg. 2008 Sep;139(3):340-7. doi: 10.1016/j.otohns.2008.05.628. PMID 18722209
- [Background] Fernandes AM, Valera FC, Anselmo-Lima WT. Mechanism of action of glucocorticoids in nasal polyposis. Braz J Otorhinolaryngol. 2008 Mar-Apr;74(2):279-83. doi: 10.1016/s1808-8694(15)31101-0. PMID 18568209
- [Background] Lee SH. Mechanisms of Glucocorticoid Action in Chronic Rhinosinusitis. Allergy Asthma Immunol Res. 2015 Nov;7(6):534-7. doi: 10.4168/aair.2015.7.6.534. Epub 2015 May 20. PMID 26333699
- [Background] Mastruzzo C, Greco LR, Nakano K, Nakano A, Palermo F, Pistorio MP, Salinaro ET, Jordana M, Dolovich J, Crimi DN, Vancheri C. Impact of intranasal budesonide on immune inflammatory responses and epithelial remodeling in chronic upper airway inflammation. J Allergy Clin Immunol. 2003 Jul;112(1):37-44. doi: 10.1067/mai.2003.1586. PMID 12847477
- [Background] Manji J, Singh G, Okpaleke C, Dadgostar A, Al-Asousi F, Amanian A, Macias-Valle L, Finkelstein A, Tacey M, Thamboo A, Javer A. Safety of long-term intranasal budesonide delivered via the mucosal atomization device for chronic rhinosinusitis. Int Forum Allergy Rhinol. 2017 May;7(5):488-493. doi: 10.1002/alr.21910. Epub 2017 Feb 2. PMID 28151588
- [Background] Palmer JN, Jacobson KW, Messina JC, Kosik-Gonzalez C, Djupesland PG, Mahmoud RA. EXHANCE-12: 1-year study of the exhalation delivery system with fluticasone (EDS-FLU) in chronic rhinosinusitis. Int Forum Allergy Rhinol. 2018 Jun 1;8(8):869-76. doi: 10.1002/alr.22141. Online ahead of print. PMID 29856520
- [Background] Thamboo A, Manji J, Szeitz A, Santos RD, Hathorn I, Gan EC, Alsaleh S, Javer AR. The safety and efficacy of short-term budesonide delivered via mucosal atomization device for chronic rhinosinusitis without nasal polyposis. Int Forum Allergy Rhinol. 2014 May;4(5):397-402. doi: 10.1002/alr.21280. Epub 2014 Jan 21. PMID 24449682
- [Background] Harvey RJ, Snidvongs K, Kalish LH, Oakley GM, Sacks R. Corticosteroid nasal irrigations are more effective than simple sprays in a randomized double-blinded placebo-controlled trial for chronic rhinosinusitis after sinus surgery. Int Forum Allergy Rhinol. 2018 Apr;8(4):461-470. doi: 10.1002/alr.22093. Epub 2018 Feb 2. PMID 29394004
- [Background] Yoo F, Ference EH, Kuan EC, Lee JT, Wang MB, Suh JD. Evaluation of patient nasal saline irrigation practices following endoscopic sinus surgery. Int Forum Allergy Rhinol. 2018 Jan;8(1):32-40. doi: 10.1002/alr.22034. Epub 2017 Oct 30. PMID 29083529
- [Background] Fox MG, Cass LM, Sykes KJ, Cummings EL, Fassas SN, Nallani R, Smith JB, Chiu AG, Villwock JA. Factors affecting adherence to intranasal treatment for allergic rhinitis: A qualitative study. Laryngoscope Investig Otolaryngol. 2022 Nov 29;8(1):40-45. doi: 10.1002/lio2.986. eCollection 2023 Feb. PMID 36846400
- [Background] Kovacs AJ, Adappa ND, Kuan EC. Exhalation Delivery Systems for Application of Intranasal Corticosteroids. Ear Nose Throat J. 2021 Jun;100(5):309-313. doi: 10.1177/0145561320980194. Epub 2020 Dec 11. PMID 33305974
- [Background] Waniewska-Leczycka M, Cieslik T, Kowalik K, Sierdzinski J, Zagor MP. Comparison of Intranasal Steroid Application Using Nasal Saline Irrigation and a Mucosal Atomization Device to Treat Chronic Rhinosinusitis. J Aerosol Med Pulm Drug Deliv. 2021 Sep;34(5):311-321. doi: 10.1089/jamp.2020.1644. Epub 2021 Apr 13. PMID 33848434
- [Background] Harvey RJ, Goddard JC, Wise SK, Schlosser RJ. Effects of endoscopic sinus surgery and delivery device on cadaver sinus irrigation. Otolaryngol Head Neck Surg. 2008 Jul;139(1):137-42. doi: 10.1016/j.otohns.2008.04.020. PMID 18585576
- [Background] Hosseini S, Wei X, Wilkins JV Jr, Fergusson CP, Mohammadi R, Vorona G, Golshahi L. In Vitro Measurement of Regional Nasal Drug Delivery with Flonase,(R) Flonase(R) Sensimist, and MAD Nasal in Anatomically Correct Nasal Airway Replicas of Pediatric and Adult Human Subjects. J Aerosol Med Pulm Drug Deliv. 2019 Dec;32(6):374-385. doi: 10.1089/jamp.2019.1523. Epub 2019 Aug 29. PMID 31464547
- [Background] Rotenberg BW. Comparison of Budesonide Delivery Via Nasal Spray and a Nasal Nebulizer to an In Vitro Adult Model. In: TP6. TP006 CLINICAL STUDIES OF ALLERGIC AIRWAY DISEASES, LUPUS, AND EOSINOPHILIC DISEASES.2021:A1338-A1338.
- [Background] NasoNeb. Particle Size and AIrflow: Implications for Nasal and Paranasal SInus Delivery. https://cdn.shopify.com/s/files/1/0373/3943/1044/files/ParticleSizeAndAirflowInNasalDrugDelivery.pdf?v=1606769959. Accessed 1/2/2025.
- [Background] Valentine R, Athanasiadis T, Thwin M, Singhal D, Weitzel EK, Wormald PJ. A prospective controlled trial of pulsed nasal nebulizer in maximally dissected cadavers. Am J Rhinol. 2008 Jul-Aug;22(4):390-4. doi: 10.2500/ajr.2008.22.3191. PMID 18702903
- [Background] Nasoneb Information for Physicians and Nurse Practitioners. Monaghan Medical Corporation. https://www.nasoneb.com/pages/physicians-nurse-practitioners. Accessed December 31, 2024.
- [Background] Manes RP, Tong L, Batra PS. Prospective evaluation of aerosol delivery by a powered nasal nebulizer in the cadaver model. Int Forum Allergy Rhinol. 2011 Sep-Oct;1(5):366-71. doi: 10.1002/alr.20057. Epub 2011 May 9. PMID 22287468
- [Background] BW R. Comparison of Budesonide Delivery Via Nasal Spray and a Nasal Nebulizer to an In Vitro Adult Model. In: TP6. TP006 CLINICAL STUDIES OF ALLERGIC AIRWAY DISEASES, LUPUS, AND EOSINOPHILIC DISEASES.2021:A1338-A1338.
- [Background] Brown K, Lane J, Silva MP, DeTineo M, Naclerio RM, Baroody FM. A pilot study of the effects of intranasal budesonide delivered by NasoNeb(R) on patients with perennial allergic rhinitis. Int Forum Allergy Rhinol. 2014 Jan;4(1):43-8. doi: 10.1002/alr.21239. PMID 24574125
- [Background] Megow A, Bouras G, Ooi EH, Vreugde S, Psaltis A, Wormald PJ. Double blind randomized controlled trial measuring the efficacy of nebulized steroid at half dose in comparison to high volume squeeze bottle steroid irrigation in management of patients with chronic rhinosinusitis. Int Forum Allergy Rhinol. 2024 Aug;14(8):1375-1377. doi: 10.1002/alr.23336. Epub 2024 Mar 13. PMID 38477174
- [Background] Wang C, Lou H, Wang X, Wang Y, Fan E, Li Y, Wang H, Bachert C, Zhang L. Effect of budesonide transnasal nebulization in patients with eosinophilic chronic rhinosinusitis with nasal polyps. J Allergy Clin Immunol. 2015 Apr;135(4):922-929.e6. doi: 10.1016/j.jaci.2014.10.018. Epub 2014 Dec 4. PMID 25483598
- [Background] Kim KT, Rabinovitch N, Uryniak T, Simpson B, O'Dowd L, Casty F. Effect of budesonide aqueous nasal spray on hypothalamic-pituitary-adrenal axis function in children with allergic rhinitis. Ann Allergy Asthma Immunol. 2004 Jul;93(1):61-7. doi: 10.1016/S1081-1206(10)61448-2. PMID 15281473
- [Background] Smith KA, French G, Mechor B, Rudmik L. Safety of long-term high-volume sinonasal budesonide irrigations for chronic rhinosinusitis. Int Forum Allergy Rhinol. 2016 Mar;6(3):228-32. doi: 10.1002/alr.21700. Epub 2016 Jan 11. PMID 26750509